CLINICAL TRIAL: NCT05122091
Title: A Single-arm, Multicenter, Open-label Phase II Study of Fruquintinib Plus SOX as a Neoadjuvant Therapy for Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Fruquintinib Plus SOX as Neoadjuvant Therapy for Locally Advanced Gastric Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Wu Liucheng, Clinical Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRUTINEOGA
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer; Fruquintinib; SOX
Keywords: Gastric cancer; Fruquintinib; Neoadjuvant; SOX
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib group (Experimental): Two-four preoperative cycles of Fruquintinib plus SOX. One cycle consists of Day 1-14 Fruquintinib 5mg oral (daily), Day 1 Oxaliplatin 130mg/M2 intravenous, Day 1-14 Tegafur gimeracil oteracil potassium capsule 40-60mg bid（dosage according to body surface area）.
  Repeated every 21st day
  Interventions: Drug: Fruquintinib + SOX

INTERVENTIONS:
Drug: Fruquintinib + SOX — Fruquintinib：5mg qd for 2 weeks on and 1 week off, q3w； SOX: Tegafur gimeracil oteracil potassium capsule: 40-60mg bid（dosage according to body surface area），d1-14，q3w； Oxaliplatin：130mg/m2，intravenous (IV) ，d1，q3w.

SUMMARY:
For locally advanced gastric/gastroesophageal junction adenocarcinoma (cT3/4aN+M0 ), neoadjuvant therapy can downstage T and N stage, improve R0 resection rate, reduce recurrence and metastasis rates, and finally improve the long-term survival. A combination of Fruquintinib and SOX for locally advanced gastric/gastroesophageal junction adenocarcinoma could be a novel therapy. This study intends to evaluate the efficacy of Fruquintinib plus SOX as neoadjuvant therapy for locally advanced gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
Gastric cancer (GC) is one of the leading causes of cancer-related deaths worldwide and a substantial global health burden. Surgery is the only possible way to cure gastric cancer, however, more than 80% of Chinese patients are diagnosed at advanced stages. Surgery and comprehensive treatment have made significant progress in gastric/gastroesophageal junction adenocarcinoma, but recurrence and metastasis are still common. Improving the R0 resection rate and reducing recurrence and metastasis rates are becoming more urgent. For locally advanced gastric/gastroesophageal junction adenocarcinoma (cT3/4aN+M0 ), neoadjuvant therapy can downstage T and N stage, improve R0 resection rate, reduce recurrence and metastasis rates, and finally improve the long-term survival. A combination of Fruquintinib and SOX for locally advanced gastric/gastroesophageal junction adenocarcinoma could be a novel therapy. This single-arm, multicenter, open-label phase II study is designed to evaluate the efficacy and safety of Fruquintinib plus SOX as neoadjuvant therapy for locally advanced gastric or gastroesophageal junction adenocarcinoma who have not received prior antitumor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ages: 18-75 Years（concluding 18 and 75 Years）;
2. Pathologically confirmed resectable or potentially resectable locally advanced gastric/gastroesophageal junction adenocarcinoma (cT3/4aN+M0) ;
3. Bone scan should be performed if bone metastasis is suspected. If peritoneal metastasis is suspected, abdominal examination should be performed to exclude distant metastasis；
4. ECOG PS 0-1, there was no deterioration within 7 days;
5. BMI≥18；
6. Has life expectancy of greater than 12 months；
7. No prior antitumor therapy (e.g., radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.)；
8. Have measurable lesions (according to RECIST 1.1);
9. The main organ functions meet the following criteria: (without blood transfusion or any blood component or cell growth factor within 14 days prior to enrollment):

   1. Absolute Neutrophil Count (ANC)≥1.5×109/L, White Blood Cell≥4.0×109/L；
   2. Platelet Count of ≥100×109/L；
   3. Hemoglobin≥90g/L；
   4. Total Bilirubin (TBIL)≤1.5 x ULN；
   5. ALT and AST≤2.5 x ULN；
   6. Urea/Urea Nitrogen（BUN）and Creatinine（Cr）≤1.5×ULN (and creatinine clearance (CCr)≥ 50mL/min);
   7. Left Ventricular Ejection Fraction (LVEF)≥50%;
   8. Electrocardiogram (ECG) Corrected QT Interval (QTcF)<470ms;
   9. INR≤1.5×ULN，APTT≤1.5×ULN;

Exclusion Criteria:

1. Received anti-VEGF/VEGFR-targeted drugs and progressed upon these drugs;
2. HER 2+;
3. Live vaccines were administered within 4 weeks prior to enrollment or possibly during the study period;
4. A history of other malignancies within 5 years prior to inclusion, except for cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery;
5. Patients with any active autoimmune disease or a documented history of autoimmune disease within 4 weeks prior to enrollment;
6. Previously received allogeneic stem cell or parenchymal organ transplantation;
7. Previously with serious cardiovascular disease, including unstable angina or myocardial infarction within 6 months prior to enrollment;
8. Known hypersensitivity to any of the study drugs or excipients;
9. Distant metastasis to any part of the body；
10. Have received other investigational treatments in clinical studies within 4 weeks prior to enrollment;
11. Any significant clinical or laboratory abnormality that the investigator considers to influence the safety evaluators;
12. Hypertension that is not controlled by the drug, and is defined as: SBP ≥150 mmHg and/or DBP ≥90 mmHg；
13. With any diseases or conditions prior to enrollment that affected drug absorption, or patients could not take drugs orally;
14. Have a gastrointestinal disease or condition that investigators suspect may affect drug absorption, including, but not limited to, active gastric and duodenal ulcers, ulcerative colitis and other digestive disease, gastrointestinal tumor with active bleeding, or other gastrointestinal conditions that may cause bleeding or perforation, according to the investigator's judgement;
15. History or presence of a serious hemorrhage (>30 ml within 3 months), hemoptysis (>5 ml blood within 4 weeks) or life threatening thromboembolic event within 12 months;
16. Have clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction; severe/unstable angina pectoris or coronary artery bypass grafting within 6 months prior to enrollment; congestive heart failure according to the New York Heart Association (NYHA) classification ≥ 2; ventricular 26 arrhythmias which needs drug treatment; or left ventricular ejection fraction (LVEF) <50%;
17. Active infection or serious infection that is not controlled by drug (≥CTCAE v5.0 Grade 2）;
18. History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×103/m); or liver cirrhosis, etc;
19. Adverse events (AEs) due to previous anti-tumor therapy has not recovered to Common Terminology Criteria for Adverse Event (CTCAE) ≤Grade 1. Alopecia, lymphocytopenia, and grade 2 neurotoxicity due to oxaliplatin are not included;
20. Women who are pregnant or lactating;
21. With blood transfusion or any blood component or cell growth factor within 14 days prior to enrollment;
22. Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions which, according to judgement of the investigator, renders the patient inappropriate for using the investigational product or affect interpretation of study results;
23. Urine routine indicates urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0 g;
24. Patients considered unsuitable for inclusion in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathological remission rate (PRR) | Approximately 2 years
  Rate of patients with < 2/3 residual tumor lesion (Grade 1b, 2, 3) in surgical specimen compared to baseline

SECONDARY OUTCOMES:
Disease free survival (DFS) | Approximately 2 years
  Disease free survival Time from randomization to relapse or death from any cause
Overall Survival (OS) | Approximately 2 years
  Overall survival Time from randomization to death from any cause
Objective response rate (ORR) | Approximately 2 years
  Rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1
Major pathological response rate (MPR) | 30 days
  Less than 10% residual carcinoma cells in the specimen
R0 resection rate | 30 days
  Evaluation of the resection margin status (positive or negative) in the rectal specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu L, Yan H, Qin Y, Huang M, Wang T, Jin Q, Wei W. Fruquintinib plus oxaliplatin combined with S-1 (SOX) as neoadjuvant therapy for locally advanced gastric cancer (GC) or gastro-oesophageal junction adenocarcinoma (GEJ): a multicentre, phase II, single-arm, open-label clinical trial (FRUTINEOGA) protocol. BMJ Open. 2024 Feb 10;14(2):e075696. doi: 10.1136/bmjopen-2023-075696. PMID 38341203